CLINICAL TRIAL: NCT00885157
Title: Immunogenicity and Safety of Fractional Booster Dose of Sanofi Pasteur's Inactivated Poliomyelitis Vaccine (IMOVAX Polio) Administered Intradermally Versus Full Booster Dose of Inactivated Poliomyelitis Vaccine (IMOVAX Polio) Administered Intramuscularly at 15 to 18 Months of Age in Healthy Toddlers in The Philippines
Brief Title: Immunogenicity and Safety of a Fractional Booster Dose of IPV Intradermally Versus Full Dose Intramuscularly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV26
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis; intradermal
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Will receive fractional doses of IPV Intradermally
  Interventions: Biological: Inactivated types 1, 2, and 3 poliovirus, D antigens
- Group B (Active Comparator): Will receive full doses of IPV Intramuscularly
  Interventions: Biological: Inactivated types 1, 2, and 3 poliovirus, D antigens

INTERVENTIONS:
Biological: Inactivated types 1, 2, and 3 poliovirus, D antigens — 0.1 mL, intradermal
  Other Names: Imovax Polio
  Arms: Group A
Biological: Inactivated types 1, 2, and 3 poliovirus, D antigens — 0.5 mL, Intramuscular
  Other Names: Imovax Polio
  Arms: Group B

SUMMARY:
The purpose of this study is to investigate the use of a fourth fractional booster dose of sanofi pasteur's IMOVAX Polio injected intradermally (using the Mantoux technique) as booster dose between 15 to 18 months of age, in terms of immunogenicity and safety.

Objectives:

* To describe in each group the immunogenicity of IMOVAX Polio administered intradermally or intramuscularly, one month after the booster dose given at 15-18 months of age in toddlers previously primed with three doses of IMOVAX Polio vaccine during the IPV25 study.
* To describe in each group the safety of the booster dose of IMOVAX Polio vaccine administered intradermally or intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 18 months on the day of inclusion
* Informed consent form signed by the parent(s) or other legally acceptable representative
* Subjects and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Child having completed all visits of the IPV25 study (NCT00604058), including the three-dose primary vaccination series with the study vaccine (IMOVAX Polio), using the route of administration as designated by randomization.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Receipt of blood or blood-derived products since birth that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine during the present trial period
* Known personal or maternal Human Immunodeficiency Virus (HIV), Hepatitis B antigen or Hepatitis C seropositivity
* History of seizures
* History of poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* Previous fourth dose vaccination against the poliomyelitis disease with either the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM injection
* Febrile illness (temperature ≥38.0 °C) or moderate or severe acute illness/infection on the day of vaccination, according to investigator judgment.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of IPV vaccine administrated intradermally as a booster vaccination. | 30 days post-vaccination
Safety: To provide information concerning the safety after booster intradermal administration of IPV vaccine | 30 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Quezon City, Manila, Philippines

REFERENCES:
- [Derived] Cadorna-Carlos J, Vidor E, Bonnet MC. Randomized controlled study of fractional doses of inactivated poliovirus vaccine administered intradermally with a needle in the Philippines. Int J Infect Dis. 2012 Feb;16(2):e110-6. doi: 10.1016/j.ijid.2011.10.002. Epub 2011 Dec 5. PMID 22153001
- See also: Related Info — http://www.sanofipasteur.com